CLINICAL TRIAL: NCT03048162
Title: The Evaluation of the Effects of Intravenous Fluids on Perfusion Index and Pleth Variability Index
Brief Title: The Effects of Intravenous Fluids on Perfusion Index and Pleth Variability Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Serkan Dogru, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OMU KAEK 2016/390
Record Dates: First submitted 2017-02-04; First posted 2017-02-09 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Perfusion
MeSH Terms: interventions — Sodium Chloride; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sodium chloride (Active Comparator): 0.9% isotonic sodium chloride, 500 ml, one package in 30 minutes
  Interventions: Drug: sodium chloride
- Hydroxyethylstarch (Active Comparator): 6% hydroxyethylstarch, 500 ml, one package in 30 minutes
  Interventions: Drug: Hydroxyethylstarch
- Ringer-Lactate Infusion Solution Bag (Active Comparator): Ringer's lactate, 500 ml, one package in 30 minutes
  Interventions: Drug: Ringer-Lactate Infusion Solution Bag

INTERVENTIONS:
Drug: sodium chloride — 500 ml of 0.9% isotonic sodium chloride
  Arms: sodium chloride
Drug: Hydroxyethylstarch — 500 ml of 6% Hydroxyethylstarch
  Arms: Hydroxyethylstarch
Drug: Ringer-Lactate Infusion Solution Bag — 500 ml of Ringer-Lactate Infusion Solution Bag
  Arms: Ringer-Lactate Infusion Solution Bag

SUMMARY:
This study is aimed to assess the effects of intravenously administered three fluid types on perfusion index and pulse variability index in patients during preoperative period. Patients will be randomly divided into three groups. Baseline, 5th, 10th, 15th, 20th, 25th and 30th min non-invasive blood pressure, oxygen saturation, heart rate, room temperature, perfusion index and pulse variability index will be measured and recorded.

DETAILED DESCRIPTION:
Intravenous volume replacement alter the dynamics of microcirculation. Perfusion index and pulse variability index are the recent parameters to evaluate the tissue microcirculatory condition. This study is aimed to assess the effects of intravenously administered three fluid types on perfusion index and pulse variability index in patients during preoperative period. Patients will be taken to recovery room in the operating theatre and wait for 15 minutes to balance the skin temperature of the patients to the environment. Patients will be randomly divided into three groups using closed envelope technique as Group L (received 500 ml of Ringer's lactate), Group S (500 ml of saline) and Group H (received 500 ml of 6% hydroxyethylstarch). Baseline, 5th, 10th, 15th, 20th, 25th and 30th min non-invasive blood pressure, oxygen saturation, heart rate, room temperature, perfusion index and pulse variability index will be measured and recorded.

ELIGIBILITY:
Inclusion Criteria:

* having a fasting period of 8 hours
* quit smoking for 8 hours before the procedure

Exclusion Criteria:

* not to participate in the study
* presence of peripheral vascular disease
* a history of upper extremity surgery
* presence of any kind of psychiatric disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Perfusion index | six months
  The perfusion of the tissues

SECONDARY OUTCOMES:
Heart rate | six months
  Heart rate
Blood pressure | six months
  Non-invasive lood pressure
Oxygen saturation | six months
  Blood oxygen saturation using pulse oximeter
Pulse variability index | six months
  The intravenous fluid requirement of the tissues

CONTACTS AND LOCATIONS:
Overall Officials: Seval Ekerer, Dr, Principal Investigator — Gaziosmanpasa University; Mustafa Suren, Dr, Principal Investigator — Gaziosmanpasa University; Serkan Karaman, Dr, Principal Investigator — Gaziosmanpasa University; Tugba Karaman, Dr, Principal Investigator — Gaziosmanpasa University; Hakan Tapar, Dr, Principal Investigator — Gaziosmanpasa University; Aynur Sahin, Dr, Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided